CLINICAL TRIAL: NCT04806061
Title: Urine Alkalinisation to Prevent AKI in COVID-19
Brief Title: Urine Alkalinisation in COVID-19
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GSTT COVID-AKI
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Covid19; Acute Kidney Injury
MeSH Terms: conditions — COVID-19; Acute Kidney Injury | interventions — Sodium Bicarbonate; Standard of Care

STUDY DESIGN:
Intervention Model Description: open label randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium bicarbonate (Experimental): iv sodium bicarbonate 8.4%
  Interventions: Drug: Sodium bicarbonate
- control (Experimental): standard care
  Interventions: Drug: standard care

INTERVENTIONS:
Drug: Sodium bicarbonate — sodium bicarbonate 8.4% to achieve urinary pH >7.5
  Other Names: sodium bicarbonate 8.4%
  Arms: sodium bicarbonate
Drug: standard care — standard care
  Other Names: usual care
  Arms: control

SUMMARY:
Since the outbreak of coronavirus disease 2019 (COVID-19), more than 100,000 patients have died in the United Kingdom. Acute kidney injury is common in critically ill patients with COVID-19. It is associated with a high risk of dying. At present, it is not clear how to prevent or treat kidney failure in these patients.

Recent research has shown that the coronavirus can directly infect kidney issue. It uses a particular protein on the cell surface (the ACE2 receptor) for entry into cells. Entry into cells is easier if the blood is more acidic.

The aim of this project is to find out whether urinary alkalisation using intravenous bicarbonate is feasible and can reduce the risk of acute kidney injury in critically ill patients with COVID-19.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is common in patients with Coronavirus disease 2019 (COVID-19). Research has shown that the SARS-CoV-2 virus can directly infect kidney issue via the Angiotensin-converting-enzyme 2 receptor which is pH dependent. The aim of this randomised controlled feasibility study is to explore whether urinary alkalisation using intravenous bicarbonate is feasible and can reduce the risk of acute kidney injury in critically ill patients with COVID-19.

Critically ill patients with COVID-19 and no AKI will be randomised to intravenous NaHCO3 8.4% versus standard care for up to 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Covid-19 positive
* Admission to Critical Care Unit
* Bladder catheter in situ
* Central line in place
* Age ≥18y
* Written informed consent to participate in the study

Exclusion Criteria:

* Stage 3 AKI (as defined by Kidney Disease Improving Global Outcome criteria)
* Chronic kidney disease stage 4 or 5
* Contraindications to NaHCO3 therapy (e.g. risk of serious drug interaction, systemic metabolic alkalosis, congestive heart failure)
* Urine pH > 7.5
* Serum sodium >150mmol/L
* Blood pressure >180/100mgHg
* Severe hypokalaemia (K<3.0mmol/L)
* Severe hypocalcaemia (Cai <0.8 mmol/L)
* Pregnant or lactating and breast-feeding women
* Patient is on a medication that may interact with sodium bicarbonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
urinary alkalisation | 10 days
  urine pH >7.5

SECONDARY OUTCOMES:
acute kidney injury | 28 days
  creatinine rise as defined by KDIGO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, PhD, Principal Investigator — Guy's & St Thomas Hospital
Locations (2):
- United Kingdom (2):
  - Guy's & St Thomas Foundation Hospital, London
  - Guy's & St Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: No